CLINICAL TRIAL: NCT01635387
Title: Upstream Use of Aliskiren in Hypertensive Haemodialysis Patients: Effects on Cardiovascular Outcomes
Brief Title: RAAS Inhibitor Drugs in Dialysis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Gennaro Cice, MD, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RAAS-block dial
Record Dates: First submitted 2012-06-27; First posted 2012-07-09 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Hypertension; End Stage Renal Disease
MeSH Terms: conditions — Hypertension; Kidney Failure, Chronic | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren (Experimental)
  Interventions: Drug: aliskiren
- Placebo (Placebo Comparator)
  Interventions: Drug: aliskiren

INTERVENTIONS:
Drug: aliskiren — 150 mg once a day per 2 week with forced uptitration to 300 mg once a day, if tolerated

SUMMARY:
Hypertensive haemodialysis patients are at high risk for cardiovascular events. This study was undertaken to ascertain whether the upstream of aliskirne, a direct renin inhibitor improves mortality and cardiovascular outcomes in these high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* chronic kidney disease stage 5
* undergoing maintenance haemodialysis for a minimum of 3 months
* existing arterial hypertension or
* history of arterial hypertension or
* resting blood pressure ≥140/90 mmHg or
* antihypertensive medication
* man and female
* 18 years and older.

Exclusion Criteria:

* recent myocardial infarction (less than 3 months)
* atrial fibrillation/atrial flutter
* hypotension with systolic blood pressure of <90 mmHg
* high-grade aortic stenosis
* left ventricular ejection fration <50%
* known allergy to aliskiren
* severe disorders of liver function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
time to first clinical event (among mortality from any cause, cardiac event including myocardial infarction, need for coronary angioplasty or coronary bypass surgery, ischaemic stroke, new-onset heart failure, new-onset atrial fibrillation) | 30 months